CLINICAL TRIAL: NCT02754219
Title: A Study to Evaluate Pharmacokinetics and Safety of Evogliptin in Subjects With Hepatic Dysfunction and Control Healthy Volunteers
Brief Title: Pharmacokinetics and Safety of Evogliptin in Subjects With Hepatic Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA1229_HI_I
Record Dates: First submitted 2016-04-27; First posted 2016-04-28 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Liver Dysfunction
Keywords: Diabetes Mellitus, Type II
MeSH Terms: conditions — Liver Diseases; Diabetes Mellitus, Type 2 | interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evogliptin (Experimental): Hepatic dysfunction, Healthy control
  Interventions: Drug: Evogliptin

INTERVENTIONS:
Drug: Evogliptin — DPP4-inhibitor, Evogliptin
  Other Names: DA-1229

SUMMARY:
The objective of the study is to compare the pharmacokinetics profiles and safety of Evogliptin in patients wit hepatic dysfunction versus healthy volunteers after single oral dose of Evogliptin

DETAILED DESCRIPTION:
When the future evogliptin be administered to liver dysfunction patients, to investgate whether dose adjustment is necessary.

ELIGIBILITY:
Inclusion Criteria:

<Hepatic Dysfunction>

* At least 6 months with chronic liver disease (Regardless of cause hepatic dysfunction)
* Child-Pugh A or B

<Healthy Control>

* Subject has the following conditions: age ± 5 years, BMI ± 20%, same sex of each matched hepatic dysfunction subject

Exclusion Criteria:

<Hepatic Dysfunction>

* Child-Pugh C
* History of Liver transplant

<Healthy Control>

* History of chronic liver disorders
* Pregnant or lactating women

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic(Cmax of Evogliptin) | Day1, Day2, Day3, Day4, Day5, Day6

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital Clinical Trial Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided